CLINICAL TRIAL: NCT04813627
Title: Epidemiological Study to Determine the Prevalence of ctDNA Positivity in Participants With Stage II (High Risk) or Stage III CRC After Surgery With Curative (R0) Intent and Subsequent Adjuvant Chemotherapy With Monitoring of ctDNA During Clinical Follow-up
Brief Title: Epidemiological Study to Monitor Study Participants With Resected Stage II (High Risk) or Stage III Colorectal Cancer for Circulating Tumor DNA Before, During and After Their Treatment With Adjuvant Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Other Study IDs: BNT000-001; DRKS00025104 (Other: Deutsches Register Klinischen Studien (German Clinical Trials Register))
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer Stage II; Colorectal Cancer Stage III
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood and tumor tissue samples collected for ctDNA assessment will be destroyed when subsequent clinical validity and/or bridging studies to support the validation of ctDNA assay are completed (where the samples are not exhausted).
  * Remaining biospecimens from a particular participant must be destroyed if the participant specifically requests that their archival specimens are destroyed upon their withdrawal from the study.
  * Remaining archival tissue blocks will be returned to the site upon request or no later than the time of final closure of the study database, whichever occurs first. For participants who are not eligible for enrollment in study BNT122-01, remaining archival tissue blocks will be returned to the site no later than 6 months after eligibility determination.
  * Remaining unused samples will be stored for a maximum of 5 years after the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with R0 resected Stage II (high risk) or Stage III CRC: The participants eligible for this epidemiological study are those with completely resected Stage II (high risk)/III CRC (per the American Joint Committee on Cancer [AJCC] 8th revised edition staging system) due to receive standard of care chemotherapy for at least 3 months following surgery.
  Interventions: Procedure: Regular blood sample collection for ctDNA assessment

INTERVENTIONS:
Procedure: Regular blood sample collection for ctDNA assessment — Blood samples for in vitro testing of ctDNA status will be drawn at study visits every 3 months for 21 months

SUMMARY:
This is a multi-site epidemiological study designed to monitor circulating tumor DNA (ctDNA) status in participants with Stage II (high risk)/III colorectal cancer (CRC) following resection/prior to adjuvant chemotherapy (AdCTx), during the course of AdCTx and for a period of up to 630 days (21 months) thereafter, according to CRC stages and disease characteristics.

Participants receive no therapeutic intervention as part of this study. This study will identify participants with confirmed Stage II (high risk)/III CRC that are positive for ctDNA after resection who might be potential candidates for the clinical study BNT122-01 (NCT04486378), a study of RO7198457 after completion of standard adjuvant chemotherapy in this patient population. These participants will have the option to enter screening for BNT122-01 at Screening Visit 2 of that study if they meet the eligibility criteria of BNT000-001 during screening. Data from the assessments from this study (BNT000-001) will be carried across to the BNT122-01 study where feasible.

DETAILED DESCRIPTION:
Individual participants will be involved in the study for at least 12 months to up to 29 months (maximum follow-up 21 months after completion of AdCTx [Visit 10]). For all participants who transfer to BNT122-01 (NCT04486378), study participation in BNT000-001 will end at time of screening for BNT122-01.

ELIGIBILITY:
Inclusion Criteria:

* Must have given informed consent indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Age ≥ 18 years old at time of signing the informed consent form.
* Ability to comply with the study protocol, in the investigator's judgment.
* Must have Stage II/Stage III rectal cancer or Stage II (high risk)/Stage III colon cancer per AJCC 2017 that has been surgically totally resected (R0 confirmed by pathology report). Stage II (high risk) colon cancer is defined as (any of):

  * T4
  * Grade ≥ 3
  * Clinical presentation with bowel obstruction or perforation
  * Histological signs of vascular, lymphatic or perineural invasion
  * < 12 nodes examined
* Adequate tumor material in formalin-fixed paraffin embedded blocks or as sectioned tissue (only upon approval by sponsor) must be available, preferably from resection. The specimen should be submitted along with an associated pathology report. Multiple samples may be provided as available, but priority should be given to tissue with the highest tumor content and lowest necrotic area.
* Intention to receive a standard of care AdCTx within 8 weeks post-surgery, and be scheduled for at least 3 months of treatment (including rest days) according to the treating physician or investigator.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Adequate end-organ function.

Exclusion Criteria:

* Neo-adjuvant (radio)chemotherapy prior to surgery.
* Prior systemic investigational therapy.
* Active Hepatitis B virus (HBV) infection.
* Active hepatitis C virus (HCV) infection.
* History of human immunodeficiency virus (HIV) antibody positivity.
* Residual tumor classification following surgery other than R0 (microscopic margin-negative resection).
* Participants with known past or current malignancy other than inclusion diagnosis, except for:

  * Cervical carcinoma of Stage 1B or less.
  * Non-invasive basal cell or squamous cell skin carcinoma.
  * Non-invasive, superficial bladder cancer.
  * Prostate cancer with a current prostate-specific antigen level < 0.1 ng/mL.
  * Any curable cancer with a complete response of > 2 years duration.
* Participant has not started standard of care AdCTx within 8 weeks post-surgery.
* Participant has received less than 3 months (including rest days) of AdCTx treatment.
* Inadequate tumor material (either quality or quantity) to support ctDNA analysis.
* Participants who have had prior splenectomy.
* Participants with diagnosed microsatellite instability high tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Stage II (high risk)/III CRC after resection (R0) and that are scheduled to receive AdCTx will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of ctDNA positivity in the post-surgery/pre-AdCTx blood sample | 4 to 8 weeks (28 to 56 days) after surgery and within 7 days prior to start of AdCTx
  Blood sample taken post-surgery and pre-adjuvant chemotherapy.

SECONDARY OUTCOMES:
Transfer of participants from the BNT000-001 study to the BNT122-01 clinical trial | 4 weeks following Visit 1 (upon availability of ctDNA positivity status)
  The absolute and relative frequency of participants that will transfer to the BNT122-01 clinical trial from this epidemiological study will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (74):
- United States (17):
  - Ridley-Tree Cancer Center, California City, California
  - John Muir Clinical Research Center, Concord, California
  - Marin Cancer Care, Greenbrae, California
  - The Oncology Institute of Hope, Los Angeles, California
  - Rocky Mountain Cancer Centers - Denver Midtown, Denver, Colorado
  - Cancer Care Specialists Of Central Illinois Sc (Ccsci) - Cancer Care Center Of Decatur, Decatur, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - USOR - New York Oncology Hematology, P.C., Albany, New York
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - USOR - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Rockwood Cancer Treatment Center, Spokane, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
- Belgium (12):
  - ZNA Campus Middelheim, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - VZW Algemeen Ziekenhuis KLINA, Brasschaat
  - Algemeen Ziekenhuis Sint-Lucas, Bruges
  - Universitair Ziekenhuis Brussel (UZ-VUB - Academisch Ziekenhuis), Jette
  - AZ Groeninge, Kortrijk
  - Centres Hospitaliers Jolimont, La Louvière
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Clinique et Maternite Sainte-Elisabeth (CMSE), Namur
  - Clinique Saint-Pierre d'ottignies (CSPO), Ottignies
  - Algemeen Ziekenhuis (AZ) Glorieux, Ronse
  - Centre Hospitalier Regional, CHR, Verviers
- Germany (29):
  - Gemeinschaftspraxis Dr. med. B. Heinrich, Prof. M. Bangerter MD, Augsburg
  - Charité Campus Mitte (CCM) - Universitätsmedizin Berlin, Berlin
  - Universitaetsklinikum St. Josef-Hospital Bochum, Bochum
  - Medizinische Klinik III, Universitätsklinikum Bonn, Bonn
  - Cancer Center Donauwoerth and Dachau, Donauwörth
  - St. Johannes Hospital, Dortmund
  - Asklepios MVZ Elmshorn, Elmshorn
  - Centrum fuer Haematologie und Onkologie Bethanien, Frankfurt am Main
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Krankenhaus Nordwest GmbH - Institut Fuer Klinisch-Onkologische Forschung, Frankfurt am Main
  - Klinikum der Johann Wolfgang Goethe-Universitaet Frankfurt, Frankfurt am Main
  - Studiengesellschaft BSF, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - Haematologisch-Onkologische Praxis Eppendorf HOPE, Hamburg
  - Asklepios Kliniken Nord, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Staedtisches Krankenhaus Kiel gGmbH, Kiel
  - Internistische Schwerpunktpraxis Hamatologie und Onkologie, Mainz
  - Ze:ro Arztpraxen, Mannheim
  - Klinikum der Universität München, Medizinische Klinik und Poliklinik III, München
  - Staedtisches Klinikum Muenchen GmbH, Klinikum Neuperlach, München
  - Prosper Hospital, Recklinghausen
  - Universitaetsmedizin Rostock, Rostock
  - Universitaetsklinikum Ulm, Ulm
  - Asklepios Klinik Weissenfels, Weißenfels
  - Helios Dr. Horst Schmidt Kliniken (HSK), Wiesbaden
  - Forschungszentrum Ruhr, Witten
- Spain (16):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Centro Oncologico Galicia, A Coruña
  - Hospital Universitari Germans Trias - ICO Badalona, Badalona
  - IOR- Instituto Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital De Sant Joan Despi Moises Broggi, Barcelona
  - Hospital General De Granollers, Granollers
  - Hospital Sant Joan de Deu-Fundacio Althaia, Manresa
  - Complejo Hospitalario de Orense, Ourense
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitari Sant Joan de Reus, Reus
  - Corporacio Sanitaria Universitaria Parc Tauli, Sabadell
  - Complejo Hospitalario Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Universitario Mutua de Terrassa, Terrassa
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No